CLINICAL TRIAL: NCT07166601
Title: An Open Label, Multicenter, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Profile of M0324, a Bispecific (MUC-1 x CD40) Antibody as Monotherapy, in Combination With Pembrolizumab, and in Combination With Chemotherapy, in Participants With Selected Advanced Solid Tumors
Brief Title: M0324 as Monotherapy and in Combination With Pembrolizumab or Chemotherapy in Participants With Selected Advanced Solid Tumors
Acronym: TITER
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS201557_0009
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor
Keywords: Bispecific CD40 agonistic antibody; Mucin-1 (MUC-1); pembrolizumab; mFOLFIRINOX; pancreatic ductal adenocarcinoma (PDAC); non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Medullary cystic kidney disease 1; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: M0324 Monotherapy (Experimental)
  Interventions: Biological: M0324
- Part 2: M0324 + Pembrolizumab (Experimental)
  Interventions: Biological: M0324; Biological: Pembrolizumab
- Part 3: M0324 + mFOLFIRINOX (Experimental)
  Interventions: Biological: M0324; Drug: mFOLFIRINOX

INTERVENTIONS:
Biological: M0324 — M0324 will be tested at increasing doses as monotherapy to determine dose-toxicity relationship and MTD (if reached) in order to support selection of recommended dose(s) for expansion (RDE).
  Arms: Part 1: M0324 Monotherapy
Biological: M0324 — M0324 will be further investigated in part 2 and part 3 of the study as combination regimen, in order to determine dose-toxicity relationship in combination and MTD (if reached) in order to support selection of RDE(s) in combination.
  Arms: Part 2: M0324 + Pembrolizumab; Part 3: M0324 + mFOLFIRINOX
Biological: Pembrolizumab — Pembrolizumab will be administered intravenously as per standard of care.
  Arms: Part 2: M0324 + Pembrolizumab
Drug: mFOLFIRINOX — mFOLFIRINOX will be administered intravenously as per standard of care.
  Arms: Part 3: M0324 + mFOLFIRINOX

SUMMARY:
The purpose of this first-in-human study is to identify a recommend dose(s) for subsequent larger studies (recommended dose(s) for expansion, RDE), examining increasing doses of M0324, primarily looking at safety, but also preliminary signs of efficacy, pharmacokinetics (PK), and pharmacodynamics (PD). Three different treatments with M0324 will be studied, M0324 as a monotherapy (Part 1), M0324 in combination with pembrolizumab (Part 2), and in combination with mFOLFIRINOX (a chemotherapy treatment) (Part 3).

ELIGIBILITY:
Inclusion Criteria:

Part 1- M0324 Monotherapy:

• Participants with certain advanced/metastatic solid tumor types known to overexpress MUC-1 and who are intolerant or refractory to standard therapy or for which no standard therapy is judged appropriate by the Investigator

Part 2- M0324 Combination with Pembrolizumab:

• Participants with certain advanced/metastatic tumor types known to overexpress MUC-1 and the participants in the combination treatment involving M0324 and pembrolizumab must be intolerant or refractory to standard therapy and no other further standard therapy should be judged appropriate by the Investigator. In addition, the participants must have had prior treatment with immune checkpoint inhibitor(s) (ICIs) and must have experienced documented disease progression on or after ICIs.

Part 3- M0324 Combination with mFOLFIRINOX:

* Participants with previously untreated metastatic pancreatic ductal adenocarcinoma, who are judged by Investigator as eligible for treatment with mFOLFIRINOX. Participants with prior Whipple surgery and/or adjuvant chemotherapy are not permitted
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Has a history of chronic diarrhea greater than or equal to (>=) Grade 2, inflammatory disease of the colon or rectum, or unresolved partial or complete intestinal obstruction
* Participant has a history of malignancy within 3 years before the date of enrollment
* Uncontrolled or poorly controlled arterial hypertension, uncontrolled cardiac arrhythmia, unstable angina, myocardial infarction, congestive heart failure [New York Heart Association (NYHA) >= II] or a coronary revascularization procedure within 180 days of study entry
* Life expectancy of less than 3 months
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2029-02-23 (Estimated); Study Completion 2029-02-23 (Estimated)

PRIMARY OUTCOMES:
Parts 1 and 2: Number of Participants With Dose Limiting Toxicities (DLTs) | Day 1 up to Day 21
Part 1, 2 and 3: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Month 40
Part 3: Number of Participants With Dose Limiting Toxicities (DLTs) | Day 1 up to Day 35

SECONDARY OUTCOMES:
Parts 1 and 2: Pharmacokinetic (PK) Plasma Concentrations of M0324 | From Day 1 up to approximately 40 months
Parts 3: Pharmacokinetic (PK) Plasma Concentrations of M0324 | From Day 1 up to approximately 40 months
Percent Change from Baseline in Pharmacodynamic Markers | From Day 1 up to approximately 40 months
  Pharmacodynamic and circulating biomarkers (e.g. cytokines) will be measured in blood.
Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator | Time from first study treatment until progressive disease or death up to approximately 40 months
Progression-Free Survival (PFS) Time Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Time from first study treatment until first documentation of progressive disease (PD) or death, assessed approximately up to 40 months
Duration of Response (DoR) According to RECIST v1.1 as Assessed by Investigator | Time from first documentation of OR until progressive disease (PD) or death, assessed approximately up to 40 months
Part 3: Overall Survival (OS) | Time from first study treatment until death, assessed approximately up to 40 months
Number of Participants With Positive Anti-Drug Antibody (ADA) of M0324 | Up to Month 40

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (5):
- United States (3):
  - Yale University School of Medicine, New Haven, Connecticut
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - NEXT Oncology, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Canada
- National Cancer Center Hospital, Chūōku, Japan

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or anew indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html